CLINICAL TRIAL: NCT06212765
Title: Effects of Oral Citrulline Supplementation on Fat-free Mass in COPD Patients With Malnutrition
Brief Title: Oral Citrulline Supplementation in COPD Patients With Malnutrition
Acronym: CITRUS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: tbp
Record Dates: First submitted 2023-12-12; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2023-10

CONDITIONS: Chronic Obstructive Pulmonary Disease Severe; Malnutrition
Keywords: COPD; L-citrulline; Malnutrition
MeSH Terms: conditions — Malnutrition; Pulmonary Disease, Chronic Obstructive | interventions — Citrulline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Citrulline (Experimental): The experimental product is 100% L-citrulline. Each pod will contain 10 grams of L-citrulline. Ten grams of L-citrulline provide 2.4 g of nitrogen.
  Interventions: Drug: L-citrulline
- Standard care (Active Comparator): The active comparator is a mixture of the six non-essential amino acids. In order for the active comparator to be iso-nitrogenated compared with the experimental product, it will provide 2.4 g of nitrogen per pod. The active comparator will combine 13.2 % alanine, 19.8 % aspartate, 11.2 % glycine, 17.1 % proline, 15.6 % serine and 23.1 % histidine, for a total of 13 g of amino acids per pod.
  Interventions: Drug: L-citrulline

INTERVENTIONS:
Drug: L-citrulline — to take 1 pod a day for 45 days

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is complicated by malnutrition in 20-70% of cases. In COPD, low fat-free mass is associated with a higher risk of morbidity and mortality. L-citrulline is a non-protein amino acid that has a direct effect on muscle protein synthesis. Oral supplementation with L-citrulline (10 g/day) in malnourished patients has shown to increase fat-free mass. The effects of L-citrulline supplementation in malnourished COPD patients are unknown.

The main objective of this prospective, single-centre, randomised, double-blind, placebo-controlled study will be to determine the impact of 45 days of nutritional supplementation with L-citrulline (10 g/day) on lean body mass (fat-free mass index (in kg.m-2) measured by bioelectrical impedance analysis) in malnourished patients (BMI < 20 kg/m2 if < 70 years old or < 22 kg/m2 if ≥ 70 years old) with COPD at stages 3-4 of the GOLD classification.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 50 and over
* COPD stage 3 or 4 according to GOLD criteria
* BMI < 20 kg/m2 if < 70 years old or < 22 kg/m2 if ≥ 70 years old
* Suspicion of sarcopenia marked by a score of 4 or more on the SARC-F questionnaire
* Absence of severe COPD exacerbation for at least 3 months

Exclusion Criteria:

* Main respiratory disease other than COPD
* Daily long-term use of systemic corticosteroids (>6 months per year, whatever the dose)
* Severe and end-stage renal insufficiency (creatinine clearance <30ml/min)
* Patient with severe hypotension, uncontrolled hypertension (at investigator's discretion)
* Contraindication to L-citrulline intake: VKA and/or cancer chemotherapy
* Osmotic diarrhoea
* Severe and/or uncontrolled progressive pathology likely to be life-threatening
* Psychiatric pathology (schizophrenia, dementia, severe bipolar/psychotic disorders, severe depressive syndrome)
* Pacemaker or other implanted electronic device

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-25 (Estimated); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-09-25 (Estimated)

PRIMARY OUTCOMES:
Fat Free Mass Index | baseline, 45+/-5 day and 1 year +/- 2 weeks
  Fat Free Mass Index (in kg.m-2) measured by bioelectrical impedance analysis

SECONDARY OUTCOMES:
Grip strength | baseline, 45+/-5 day and 1 year +/- 2 weeks
  Grip strength will be measured using a dynamometer with the patient in a seated position, elbow bent at 90°, shoulders relaxed and forearm in a neutral position. The dynamometer should be held in the dominant hand. The measurement should be taken twice. The highest value will be used.
Maximum quadriceps strength | baseline, 45+/-5 day and 1 year +/- 2 weeks
  The maximum voluntary force of the quadriceps of the left lower limb will be measured on a weight bench using a strain gauge to determine force during isometric contraction (at 90° knee flexion). The position of the patient will be standardized: arms crossed over the chest, no back support during the measurement and no support of the hips and contralateral leg to avoid any compensatory movement. Three reproducible measurements (+/-10%) will be taken at 1 min intervals, with the highest value selected.
6-minute walk test | baseline, 45+/-5 day and 1 year +/- 2 weeks
  The 6-min walking test (6MWT) measures the distance that a patient can walk on an indoor 30-m flat corridor for a 6-min period. Due to a familiarisation effect, two tests will be performed, with at least 15 min of intervening rest, with the greatest distance in the two tests being recorded. The 6-min walking distance (6MWD) will be expressed in metres. Other variables will be measured: minimum pulse oxygen saturation (SpO2), peak heart rate and dyspnoea and fatigue ratings at the end of test.
Quality of life questionnaires | baseline, 45+/-5 day and 1 year +/- 2 weeks
Number of steps walked daily measured by actigraphy | baseline, 45+/-5 day and 1 year +/- 2 weeks
  Actigraphy is an objective measurement of physical activity using a device that measures acceleration and movement (accelerometer). The number of steps walked daily is used to assess free daily-living activity in clinical trials. It is measured using an accelerometer worn 24 hours a day during five days. In this study, we will use the triaxial accelerometer Actigraph GT3X®. Instructions for the medical device use are provided on the website https://www.theactigraph.com.
  The patient will be instructed to wear the accelerometer around the wrist 24 hours a day during 5 consecutive days including week-end and will be asked to maintain usual routine activity. The number of steps walked daily will be the average of the daily number of steps over the five days.
Flow-mediated dilation | baseline, 45+/-5 day and 1 year +/- 2 weeks
  Flow-mediated dilatation (FMD) of the brachial artery will be calculated according to standard recommendations. Briefly, a pneumatic cuff will be placed on the right forearm distal to the elbow. The probe will be placed approximately midway between the antecubital and axillary regions and secured with a stereoscopic arm. Basal diameter and velocity will be recorded continuously for a minimum period of one minute. The cuff will then be inflated to 250 mm Hg for 5 minutes before sudden deflation to induce post-ischemic hyperemia. Fifteen minutes later, baseline measurements will be repeated to measure endothelial-independent, nitrate-induced dilatation. Nitrate-induced dilatation (NMD) will be calculated 4 min after sublingual administration of 0.3 mg trinitrin (NATISPRAY, Teofarma S.R.L. Italy). FMD and NMD will be expressed as a percentage change in basal diameter and in mm, after post-ischemic hyperemia and after administration of nitrate derivatives, respectively.
BODE index | baseline, 45+/-5 day and 1 year +/- 2 weeks
  The BODE index is a multidimensional index of disease severity in COPD that incorporates four independent predictors: the body mass index (BMI), the degree of airflow obstruction assessed by the Forced Expiratory Volume in one second (FEV1), the modified Medical Research Council (mMRC) dyspnea scale, and the exercise capacity assessed by the 6-min walking distance (6MWD) test.
COPD Assessment Test (CAT) | baseline, 45+/-5 day and 1 year +/- 2 weeks
  the COPD Assessment Test (CAT) is a patient-completed questionnaire assessing globally the impact of COPD (cough, sputum, dysnea, chest tighteness) on health status. CAT scores range from 0 to 40. Higher scores indicate a more severe impact of COPD on the patient's life. The difference between stable and exacerbating patients is five units. No target score represents the best possible outcome.
Visual Simplified Respiratory Questionnaire (VSRQ) | baseline, 45+/-5 day and 1 year +/- 2 weeks
  The Visual Simplified Respiratory Questionnaire (VSRQ) is designed to assess health-related quality of life (HRQoL) in patients with chronic obstructive pulmonary disease (COPD). It contains eight items: dyspnea, anxiety, depressed mood, sleep, energy, daily activities, social activities and sexual life.
mMRC dyspnea scale | baseline, 45+/-5 day and 1 year +/- 2 weeks
  the Modified Medical Research Council (mMRC) Dyspnea Scale Stratifies severity of dyspnea in respiratory diseases, particularly COPD. The higher the degree, the more severe the shortness of breath.
DIsability RElated to COPD Tool (DIRECT) | baseline, 45+/-5 day and 1 year +/- 2 weeks
  The DIsability RElated to COPD Tool (DIRECT) is a 10-item questionnaire that specifically assesses COPD-related disability.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: when all the data has been analysed and published